CLINICAL TRIAL: NCT01774071
Title: A Phase I/II Study of 89Zr-DFO-MSTP2109A in Patients With Prostate Cancer
Brief Title: Study of 89Zr-DFO-MSTP2109A in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-178
Record Dates: First submitted 2013-01-11; First posted 2013-01-23 (Estimated); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: 89Zr-DFO-MSTP2109A; tracer; pet scan; 12-178
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (2):
- 89Zr DFOMSTP2109A tracer Group 1 (Experimental): The first group of participants will include 6 participants whom will receive 10mg of 89Zr-DFO-MSTP2109A. A second group of 6 participants may receive twice the amount of antibody to determine if this results in better pictures of your tumors. Once we determine whether 10 mg or the larger 20 mg dose of 89Zr-DFOMSTP2109A is best and well tolerated we will use that amount for future participants in Group 2.
  Interventions: Drug: 89Zr- DFO-MSTP2109A
- 89Zr-DFO-MSTP2109A tracer Group 2 (Experimental): Once we determine whether 10 mg or the larger 20 mg dose of 89Zr-DFOMSTP2109A is best and well tolerated we will use that amount for future participants in Group 2. Group 2 will include up to 15 participants whom may receive a dose of up to 20mg.
  Interventions: Drug: 89Zr DFO-MSTP2109A

INTERVENTIONS:
Drug: 89Zr- DFO-MSTP2109A — If you are enrolled onto Group 1:
  Once you are given the diagnostic agent, the following procedures will be done:
  PET scans at the approximate times:
  * 1-4 hours after the injection
  * 24 hours after the injection (the next day, Day 2)
  * 48-120 hours after the injection (on either Day 3, 4, or 5)
  * 144-168 hours after the injection (on either Day 6, 7, or 8) You will also have research bloods drawn on the following times and days,
  * Day 1: before the injection, approximately 5 minutes after, 30 minutes after, 1 hour after and 2-4 hours after the injection.
  * At each time of your scheduled PET scan.
  Arms: 89Zr DFOMSTP2109A tracer Group 1
Drug: 89Zr DFO-MSTP2109A — If you are enrolled onto Group 2:
  Once you are given the study drug, the following procedures will be done:
  You will have one PET scan done. The timing of the PET scan will be determined at the time of your enrollment (~ 3-7 days after injection).
  No research blood work will be drawn in Group 2
  Arms: 89Zr-DFO-MSTP2109A tracer Group 2

SUMMARY:
The purpose of this study is to see if a new diagnostic research agent named 89Zr-DFO-MSTP2109A can show prostate cancer tumors on a PET scan; as well as see how long 89Zr-DFO-MSTP2109A lasts in the blood when given in small amounts. DFO-MSTP2109A is an antibody that works against STEAP1 - found on the surface of prostate cancer cells. Attached to the DFO-MSTP2109A is a radioactive material called 89ZR, which allows it to be imaged by a PET scanner. The results of this study may help researchers know whether 89Zr-DFO-MSTP2109A can be used as a diagnostic agent for finding prostate cancer that have STEAP1 on its surface with a PET scanner. The reason why identifying STEAP1 on prostate cancer cells is that new therapies are being developed to target STEAP1 prostate cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study, patients should be eligible for enrollment into protocol 11-016 (therapy with the DSTP3086S ADC) or meet all of the following criteria:
* Patients meeting the criteria for enrollment on research protocol 11-016 to receive DSTP3086S ADC (therapeutic ADC based on MSTP2109A) will be the preferred patients for this study. Patients that are to receive DSTP3086S will not be injected with DSTP2086S until imaging with 89Zr-DFOMSTP2109A is finished, approximately 1 week.
* Adult male > 21years of age
* Visible lesions by either CT, bone scan or MRI consistent with metastatic disease
* Metastatic progressive disease
* Imaging modalities:
* Bone scan: new osseous lesion and/or MRI or CT: An increase in measurable soft tissue disease or the appearance of new sites of disease.

Or

* PSA changes over range of value 26%
* Patients with histologically confirmed prostate cancer at MSKCC
* STEAP1 antigen positive tissue known from prior IHC testing or if STEAP1 status is not known archival sample will be sent to Genentech for IHC. Samples need to be positive, when feasible metastatic lesions will be tested preferentially rather than the primary.
* Performance status of 60 or higher (Karnofsky scale) (Appendix A)
* Ability to understand and willingness to sign a written informed consent document
* PSA levels to be taken within 2 weeks of antibody administration.

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria will not be eligible for study entry:
* Previous anaphylactic reaction to human, humanized or chimeric antibody
* Hematologic
* Platelets <75K/mcL
* ANC <1.0 K/mcL
* Hepatic laboratory values
* AST/ALT >2.5 x ULN
* Renal laboratory values
* Bilirubin >1.5 x ULN (institutional upper limits of normal)
* eGFR < 30mL/min/1.73m2
* Patients with history of hypersensitivity reaction to any component of 89Zr-DFOMSTP2109A, including DFO

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-01; Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Larson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Martiniova L, Zielinski RJ, Lin M, DePalatis L, Ravizzini GC. The Role of Radiolabeled Monoclonal Antibodies in Cancer Imaging and ADC Treatment. Cancer J. 2022 Nov-Dec 01;28(6):446-453. doi: 10.1097/PPO.0000000000000625. PMID 36383907
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- 89Zr DFOMSTP2109A Tracer Group 1 - 10mg: The first group of participants will include 6 participants whom will receive 10mg of 89Zr-DFO-MSTP2109A. A second group of 6 participants may receive twice the amount of antibody to determine if this results in better pictures of your tumors. Once we determine whether 10 mg or the larger 20 mg dose of 89Zr-DFOMSTP2109A is best and well tolerated we will use that amount for future participants in Group 2.
  89Zr- DFO-MSTP2109A: If you are enrolled onto Group 1:
  Once you are given the diagnostic agent, the following procedures will be done:
  PET scans at the approximate times:
  * 1-4 hours after the injection
  * 24 hours after the injection (the next day, Day 2)
  * 48-120 hours after the injection (on either Day 3, 4, or 5)
  * 144-168 hours after the injection (on either Day 6, 7, or 8) You will also have research bloods drawn on the following times and days,
  * Day 1: before the injection, approximately 5 minutes after, 30 minutes after, 1 hour after and 2-4 hours after the injection.
  * At each time of your scheduled PET scan.
- 89Zr-DFO-MSTP2109A Tracer Group 2: Once we determine whether 10 mg or the larger 20 mg dose of 89Zr-DFOMSTP2109A is best and well tolerated we will use that amount for future participants in Group 2. Group 2 will include up to 15 participants whom may receive a dose of up to 20mg.
  89Zr DFO-MSTP2109A: If you are enrolled onto Group 2:
  Once you are given the study drug, the following procedures will be done:
  You will have one PET scan done. The timing of the PET scan will be determined at the time of your enrollment (~ 3-7 days after injection).
  No research blood work will be drawn in Group 2
Period: Overall Study
Arm/Group | 89Zr DFOMSTP2109A Tracer Group 1 - 10mg | 89Zr-DFO-MSTP2109A Tracer Group 2
Started | 19 | 0
Completed | 19 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants recruited for Group 2
Groups:
- 89Zr DFOMSTP2109A Tracer Group 1: The first group of participants will include 6 participants whom will receive 10mg of 89Zr-DFO-MSTP2109A. A second group of 6 participants may receive twice the amount of antibody to determine if this results in better pictures of your tumors. Once we determine whether 10 mg or the larger 20 mg dose of 89Zr-DFOMSTP2109A is best and well tolerated we will use that amount for future participants in Group 2.
  89Zr- DFO-MSTP2109A: If you are enrolled onto Group 1:
  Once you are given the diagnostic agent, the following procedures will be done:
  PET scans at the approximate times:
  * 1-4 hours after the injection
  * 24 hours after the injection (the next day, Day 2)
  * 48-120 hours after the injection (on either Day 3, 4, or 5)
  * 144-168 hours after the injection (on either Day 6, 7, or 8) You will also have research bloods drawn on the following times and days,
  * Day 1: before the injection, approximately 5 minutes after, 30 minutes after, 1 hour after and 2-4 hours after the injection.
  * At each time of your scheduled PET scan.
- Total: Total of all reporting groups
Arm/Group | 89Zr DFOMSTP2109A Tracer Group 1 | 89Zr-DFO-MSTP2109A Tracer Group 2 | Total
Number analyzed (Participants) | 19 | 0 | 19
Age, Continuous [Median (Full Range); unit: years] | 66 [48 to 80] |  | 66 [48 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 19 |  | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 18 |  | 18
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 19 |  | 19
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 |  | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Histologically Positive Lesions That Are Positive on Imaging
Description: Antibody imaging will be considered feasible if 75% of the patients are antibody-imaging-positive. We will enroll 6 patients (cohort 1A) at the 10mg dose level for an initial decision on feasibility. If 4 or more of these patients have 20% or more of their active lesions detectable by 89Zr-DFO-MSTP2109A then we will consider the agent feasible for imaging, otherwise we will proceed to cohort 1B. If the true feasibility rate is 40%, this rule will affords more than 82% chance that cohort 1B will be opened for enrollment; this probability is less than 17% if the true feasibility is 75%.
Time Frame: 2 years
Population: Participants not enrolled into Group 2
Measure: Number (95% Confidence Interval); unit: % of participants with + lesions
Arm/Group | 89Zr DFOMSTP2109A Tracer Group 1 | 89Zr-DFO-MSTP2109A Tracer Group 2
Number analyzed (Participants) | 19 | 0
% of participants with + lesions | 86 [75 to 100] |

2. Primary Outcome: Number of Participants Evaluated for AEs
Description: All participants will be evaluated for adverse events which will be graded for intensity on a scale of 0 to 5. Severity grades will be recorded and based on the CTCAE v4.0. Adverse events will be defined graded using CTCAE V4.0.
Time Frame: 2 years
Population: Participants not enrolled into Group 2
Measure: Count of Participants; unit: Participants
Arm/Group | 89Zr DFOMSTP2109A Tracer Group 1 | 89Zr-DFO-MSTP2109A Tracer Group 2
Number analyzed (Participants) | 19 | 0
Participants | 19 |

3. Primary Outcome: Rate of Clearance of Tracer 89Zr-DFO-MSTP2109A
Description: Serial blood draws will be used to estimate the pharmacokinetic profile of the 10mg 89Zr-DFO-MSTP2109A in this patient population. Blood samples will be obtained in green top tube: Just prior to injection of 89Zr-DFO-MSTP2109A (baseline)Approximately 5 ± 2, 15 ± 5, 30 ± 9, 60 ± 19, and 120 to 240 minutes after injection of the tracer. One sample at the time of each subsequent day of imaging (24 + 8h, ~48-96h and ~120-168h post injection).
Time Frame: up to 168 hours
Population: Participants not enrolled to Group 2
Measure: Median (Full Range); unit: mL/hour
Arm/Group | 89Zr DFOMSTP2109A Tracer Group 1 | 89Zr-DFO-MSTP2109A Tracer Group 2
Number analyzed (Participants) | 19 | 0
mL/hour | 19.7 [0.64 to 79.7] |

4. Primary Outcome: Biodistribution/SUVmax
Description: A PET-CT scan extending from top of skull to mid thighs will be performed to determine the biodistribution/SUVmax in bone and soft tissue
Time Frame: 2 years
Population: Participants not enrolled to Group 2
Measure: Median (Full Range); unit: g/mL
Arm/Group | 89Zr DFOMSTP2109A Tracer Group 1 | 89Zr-DFO-MSTP2109A Tracer Group 2
Number analyzed (Participants) | 19 | 0
g/mL
  SUVmax in bone | 20.6 [4.4 to 59.3] |
  SUVmax in soft tissue | 16.8 [9.0 to 24.0] |

5. Secondary Outcome: Percentage of Histologically Positive Lesions That Were True Positive on PET Imaging
Description: Ability of 89Zr-DFO-MSTP2109A PET to detect sites of metastatic prostate cancer.
Time Frame: 2 years
Population: Participants not enrolled in Group 2
Measure: Number (95% Confidence Interval); unit: % of positive lesions
Units Other Than Participants: lesions
Arm/Group | 89Zr DFOMSTP2109A Tracer Group 1 | 89Zr-DFO-MSTP2109A Tracer Group 2
Number analyzed (Participants) | 19 | 0
Number analyzed (lesions) | 17 | 0
% of positive lesions | 86 [75 to 100] |

ADVERSE EVENTS:
Time Frame: 2 years
Description: Participants not enrolled to Group 2
Arm/Group | 89Zr DFOMSTP2109A Tracer Group 1 | 89Zr-DFO-MSTP2109A Tracer Group 2
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/0
Other Adverse Events (participants affected / at risk) | 0/19 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT01774071/Prot_SAP_000.pdf